CLINICAL TRIAL: NCT00396955
Title: A Multicenter, Randomized, Double-Blind Comparison of 4 Dose Regimens of Pla-695, Naproxen, and Placebo Administered Daily for 6 Weeks in Subjects With Active Osteoarthritis of the Knee
Brief Title: A Study Comparing 4 Dose Regimens of PLA-695, Naproxen, and Placebo In Subjects With Osteoarthritis Of The Knee
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: imbalance of gastrointestinal and the lipase events
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3175A1-202
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; arthritis; pain
MeSH Terms: conditions — Osteoarthritis; Arthritis; Pain | interventions — PLA-695

INTERVENTIONS:
Drug: PLA-695

SUMMARY:
Objectives: Primary:To assess the efficacy and safety of PLA-695 in subjects with active osteoarthritis (OA) of the knee.

Secondary:To determine the pharmacokinetics (PK) and pharmacodynamics (PD) of PLA-695 among dose levels. To assess health outcome measures. To assess the effect of PLA-695 on biomarkers related to clinical responses. To assess PLA-695 exposure-response relationship on PD, efficacy, and safety measures. To assess pharmacogenomics (PGX) analysis in OA.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, double-dummy, parallel, placebo- and positive-control (naproxen), dose-ranging study to assess the efficacy and safety of 3 oral doses of PLA-695 administered QD and 1 dose of PLA-695 administered BID for 6 weeks. Subjects will be randomized to 1 of 6 treatment groups: PLA-695 50 mg, 200 mg, or 400 mg QD, PLA-695 200 mg BID, placebo, or naproxen 500 mg BID. Subjects will undergo a washout period of 2 to 14 days. The number of days for washout will be determined by the pre-study NSAID of each subject. Subjects who washout from previous therapy with an increase in signs and symptoms of OA will be randomly assigned to receive PLA-695.

ELIGIBILITY:
Inclusion Criteria: The main inclusion criteria is listed below, additional inclusion criteria is in the protocol.

* Men or women 50 to 75 years of age. Women must be of non-childbearing potential. Sexually active men who are not surgically sterile must agree and commit to use of barrier contraception during the study and for at least 12 weeks after the last dose of PLA.
* Diagnosed with idiopathic OA of the knee for at least 3 months duration in accordance with [1986] American College of Rheumatology (ACR) clinical and radiographic criteria: knee pain, the presence of osteophytes, and any one of the following: age >50 years, crepitus, or morning stiffness <30 minutes.
* Radiographic confirmation of OA at the target joint (weight-bearing anteroposterior and lateral views) within 1 year of screening.
* Must be currently treated for OA with a stable daily dose of 1 NSAID, including COX-2 inhibitors, not exceeding the maximum recommended dose in the product label, and taken as prescribed by the physician, starting at least 4 weeks before the screening visit.

Exclusion Criteria: These are some of the main exclusion criteria for the the study. Additional exclusion are included in the protocol.

* History of or suspected current esophageal or gastrointestinal bleeding, ulcers, obstruction, or perforation, or pancreatitis.
* Grade 4 severity on the Kellgren-Lawrence Scale on the screening target knee radiograph.
* Any significant cardiovascular, hematologic, blood dyscrasia, endocrine, respiratory, neurologic, psychiatric, metabolic, immunologic, infectious, hepatic, or renal condition that the investigator considers detrimental to the subject's participating in the study or that may prevent the successful completion of the study.
* Any clinically significant laboratory abnormality.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
WOMAC VAS walking pain (question 1) at week 6 is the primary endpoint.

SECONDARY OUTCOMES:
WOMAC VAS walking pain at weeks 1, 2, 3, 4, and 5; WOMAC pain, stiffness, and function subscales, and composite score; Investigatorsâ Efficacy Evaluation; Investigatorsâ overall assessment; Joint tenderness. Subjectsâ Efficacy Evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Argentina, Scheima@wyeth.com; Trial Manager, Principal Investigator — For Brazil, xavierl@wyeth.com; Trial Manager, Principal Investigator — For China, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Hong Kong, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Hungary, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For Mexico, gomezzlj@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Spain, infomed@wyeth.com
Locations (77):
- United States (37):
  - Huntsville, Alabama
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Palo Alto, California
  - Rancho Mirage, California
  - Santa Maria, California
  - Upland, California
  - Delray Beach, Florida
  - Fort Lauderdale, Florida
  - Ocala, Florida
  - Palm Harbor, Florida
  - South Miami, Florida
  - Tampa, Florida
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Wichita, Kansas
  - Baltimore, Maryland
  - Frederick, Maryland
  - Fall River, Massachusetts
  - Kalamazoo, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Dover, New Hampshire
  - Mamaroneck, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Duncansville, Pennsylvania
  - West Reading, Pennsylvania
  - Willow Grove, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin
- Argentina (3):
  - Capital Federal, Buenos Aires
  - Cordoba-Capital, Córdoba Province
  - San Miguel de Tucumán, Tucumán Province
- São Paulo, São Paulo, Brazil
- Canada (15):
  - Coquitlam, British Columbia
  - Kelowna, British Columbia
  - Langley, British Columbia
  - Penticton, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Trois-Rivières, Quebec
- Hong Kong, Hong Kong
- Hungary (5):
  - Békéscsaba
  - Budapest
  - Debrecen
  - Kiskunhalas
  - Nyíregyháza
- Mexico (3):
  - Guadalajara, Jalisco
  - Monterrey, Nuevo León
  - Mexico City
- Netherlands (4):
  - 's-Hertogenbosch
  - Almere Stad
  - Geleen
  - Nijmegen
- Poland (4):
  - Krakow
  - Szczecin
  - Warsaw
  - Wroclaw
- Spain (4):
  - A Coruña
  - Guadalajara
  - Madrid
  - Seville